CLINICAL TRIAL: NCT02171312
Title: Clinical Evaluation of a Novel Balance, Vestibular and Oculomotor Assessment Tool
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency); National Football League (Other); General Electric (Industry); UnderArmour (Unknown)
Responsible Party: Principal Investigator, David Wright, Associate Professor, Emory University
Other Study IDs: IRB00075343
Record Dates: First submitted 2014-06-19; First posted 2014-06-24 (Estimated); Last update posted 2016-02-09 (Estimated); Status verified 2015-10

CONDITIONS: Mild Concussion; Post Concussion Syndrome; Vestibular Neuritis
Keywords: Dizziness; Imbalance
MeSH Terms: conditions — Brain Concussion; Post-Concussion Syndrome; Vestibular Neuronitis; Dizziness

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Concussion Cohort: Participants with possible concussion related dizziness will complete iDETECT battery testing and routine balance and vestibular testing.
  Interventions: Device: iDETECT Assessment; Behavioral: Routine Balance and Vestibular Testing
- Healthy Controls: Participants without possible concussion related dizziness will complete iDETECT battery testing and routine balance and vestibular testing.
  Interventions: Device: iDETECT Assessment; Behavioral: Routine Balance and Vestibular Testing

INTERVENTIONS:
Device: iDETECT Assessment — The iDETECT device is an open platform for an evaluation of cognitive, balance, and oculomotor performance after mild traumatic brain injury (mTBI). It is a rugged, portable, neurocognitive assessment tool designed specifically for use in field and triage settings for the rapid evaluation of functional neurologic impairment after potential concussive injury. The apparatus includes an enhanced heads-up display visor with integration motion detection technology, noise-reducing headphones optimized with pink noise, and a handheld display for test battery administration, subject response inputs, and user data output. iDETECT will be used to assess multimodal neurologic function in participants.
  Other Names: integrated Display Enhanced Testing for Cognitive Impairment and mild traumatic brain injury (iDETECT)
Behavioral: Routine Balance and Vestibular Testing — A clinician will assess balance and vision by standard of care routine tests for neurologic function.

SUMMARY:
The iDETECT (Integrated Display Enhanced Testing for Concussion and mild traumatic brain injury) system is a novel portable, open access platform that enables immediate and rapid assessment of multimodal neurologic function. This study seeks to evaluate the iDETECT function testing battery with currently used balance and inner ear assessment methods during initial concussion clinic referral. Two groups of participants will be enrolled; a concussion related dizziness cohort and control subjects. The investigators will enroll the concussion cohort from patients presenting to the Sports Concussion Institute (SCI) with persistent dizziness and imbalance symptoms following possible concussion. Healthy control participants will be recruited from the local community. iDETECT's ability to identify post concussion balance/vestibular disturbances will be compared to an expert concussion assessment. Both cohorts will participate in the iDETECT assessment and the clinical assessment.

DETAILED DESCRIPTION:
The iDETECT (Integrated Display Enhanced Testing for Concussion and mild traumatic brain injury) system is a novel portable, open access platform that enables immediate and rapid assessment of multimodal neurologic function. This study seeks to evaluate and validate the iDETECT balance, vestibular, and oculomotor testing battery with clinician performed balance and vestibular assessment methods. Two groups of participants will be enrolled; concussion related dizziness cohort and control subjects (no concussion or dizzy symptoms). The investigators will enroll the concussion cohort from patients presenting to the Sports Concussion Institute (SCI) with persistent dizziness and imbalance symptoms following possible concussion. Healthy control participants with normal vestibular function and no history of concussion will be recruited from the local community. All participants will be tested with both the iDETECT balance and vestibular assessment battery and the current clinical reference standards for imbalance and vestibular dysfunction performed by a clinician. Performance on the iDETECT balance and vestibular assessment battery will be compared between normal controls and the concussion cohort.

ELIGIBILITY:
Concussion Cohort

Inclusion Criteria:

* Age ≥ 12
* History of concussion within prior 6 months
* Complaint or symptoms of dizziness / balance problems

Exclusion Criteria:

* History of any of the following:Depression, sleep apnea, seizure disorder, migraine headaches, prior brain or spine surgery, peripheral neuropathy, lower extremity orthopedic problems
* Chronic drug or alcohol use; or drug or alcohol use within the previous 24 hours.

Control Cohort

Inclusion Criteria:

* Age ≥ 12
* Physically active (at least 60 min of exercise, team-based or recreational, 3 times of week)

Exclusion Criteria:

* Concussion or concussive-like symptoms within prior 6 months
* Current complaint or symptoms of dizziness/balance problems
* History of any of the following:

Depression, sleep apnea, seizure disorder, claustrophobia, prior central nervous system (CNS) surgery, peripheral neuropathy, developmental delay, learning disabilities lower extremity orthopedic problems that prevent standing or walking

* Participants also cannot currently be the under care of a doctor these or any related conditions that may cause cognitive impairment.
* Chronic drug or alcohol use; or drug or alcohol use within the previous 24 hours

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: A cohort of patients presenting to the Sports Concussion Institute with persistent post concussive dizziness and imbalance will be enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2015-04; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Simulator Sickness assessed by the Simulator Sickness Questionnaire (SSQ) | Post iDETECT testing (Up to three minutes)
  The Simulator Sickness Questionnaire (SSQ) is a 16-item simulator sickness questionnaire. Participants mark the extent to which they are experiencing various after effects on a scale from 0 to 3 with higher numbers indicating greater severity.
Presence of Post Concussive Symptoms assessed by the Post Concussion Symptoms Scale (PCSS) | Post iDETECT testing (Up to three minutes)
  The Post Concussion Symptoms Scale (PCSS) is a self-report measure with 22 post concussive symptom items graded on a scale from 0 (no symptoms) to 6 (severe symptoms).
User Experience assessed by the iDETECT User Experience Survey | Post iDETECT testing (Up to three minutes)
  The iDETECT User Experience Survey will be used to evaluate participant's experiences with iDETECT as is designed to gather information to help investigators improve the design and effectiveness of iDETECT. It is a thirteen point questionnaire in which participants will rate their experience with the iDETECT tool on a scale from "strongly agree" and "strongly disagree".

SECONDARY OUTCOMES:
Imbalance assessed by the Balance Error Scoring System (BESS) Score | Visit 0 (Up to ten minutes)
  The Balance Error Scoring System (BESS) is a quantitative measure of balance designed for evaluation of imbalance following sports concussion. The BESS is organized into a series of 6 conditions of increasing difficulty. Subjects perform a series of three stances for 20 seconds each standing on either a hard surface or a soft foam surface. Subjects are examined in these six separate conditions with eyes closed. The six balance conditions are; (1) double leg stance, hard surface; (2) single leg stance, hard surface; (3) tandem stance, hard surface; (4) double leg stance, foam surface; (5) single leg stance, foam surface; (6) tandem stance, foam surface. An examiner scores each condition with zero errors representing perfect balance and a maximum of 10 scored errors for each balance condition. The overall score is a composite balance score ranging from zero errors to a maximum score of 60 errors with lower scores representing better balance.
Postural Stability assessed by Quantitative Balance Testing (BioSway) Score | Visit 0 (Up to five minutes)
  Quantitative Balance Testing (BioSway) provides information about postural stability by measuring subjects sway on a force platform under different conditions. Tests of sensory organization are used to evaluate sensory and postural responses using a series of conditions of increased difficulty.Subjects stand on a force platform that estimates sway in a horizontal antero-posterior direction. Subjects are examined in four separate conditions; (1) eyes open, fixed surface. (2) eyes closed, fixed surface; (3) eyes open, foam surface; (4) eyes closed, foam surface. Each condition is scored according to sway, where 100 is no sway and 0 is a subject fall.
Visual Acuity assessed by the Dynamic Visual Acuity (DVA) Test | Visit 0 (Up to five minutes)
  Dynamic Visual Acuity (DVA) is a measure of visual acuity during head movement using customized computerized software. Visual acuity during head movement will be measured using a computerized system in which subjects read screen based characters while performing horizontal head movements at a target head velocity is between 120 - 180°/sec.
Vestibular Function assessed by Vestibular/Ocular-Motor Screening (VOMS) | Visit 0 (Up to ten minutes)
  The Vestibular/Ocular-Motor Screening (VOMS) is a quantitative measure of vestibular function assessing subjective symptoms when subjects perform a variety of vestibular and oculomotor tasks. VOMS includes symptoms assessments during smooth pursuit, saccades, horizontal and vertical vestibular ocular reflex, near point convergence, and a visual motion sensitivity test.
Dynamic Gait Ability assessed by Dynamic Gait Index (DGI) Score | Visit 0 (Up to ten minutes)
  The Dynamic Gait Index (DGI) is used to measure dynamic gait stability and fall risk. Scoring of the DGI is based on a 4- point scale from 0 (severe impairment) to 3 (normal ability). A maximum total score of 24 is possible and scores less than 20 indicate fall risk.
High Level Balance assessed by the High-level Mobility Assessment Tool (HiMAT) | Visit 0 (Up to ten minutes)
  The High-level Mobility Assessment Tool (HiMAT) is used assess high-level balance designed specifically to address the ceiling effect in traumatic brain injury outcome measures. Scoring of the HiMAT is based on performance on eight, timed mobility tasks scored on a 4-point scale with increasing scores representing poor performance on each task. A maximum total score of 32 is possible.
Mobility assessed by the High-level Mobility Assessment Tool (HiMAT) | Visit 0 (Up to ten minutes)
  The High-level Mobility Assessment Tool (HiMAT) is used assess mobility designed specifically to address the ceiling effect in traumatic brain injury outcome measures. Scoring of the HiMAT is based on performance on eight, timed mobility tasks scored on a 4-point scale with increasing scores representing poor performance on each task. A maximum total score of 32 is possible.
Confidence in Balance assessed by the Activities-specific Balance Confidence (ABC) Scale | Visit 0 (Up to ten minutes)
  The Activities-specific Balance Confidence (ABC) Scale is used to measure confidence in balance across a continuum of 16 activities including progressively challenging situations from mobility in the home to walking on icy sidewalks.Total scores range from 0 - 100% with baseline scores of < 80% considered abnormal. A significant change in the ABC score is either a return to a score of at least 80% or a change of more than 10 points.
Dizziness assessed by the Dizziness Handicap Inventory (DHI) | Visit 0 (Up to ten minutes)
  The Dizziness Handicap Inventory (DHI) is a 25-item self-assessment inventory designed to evaluate the self-perceived effects of dizziness. Total scores range from 0 - 100 with higher scores reflecting greater perceived handicap due to dizziness.
Visual Vertigo Symptoms assessed by the Visual Vertigo Analog Scale (VVAS) | Visit 0 (Up to ten minutes)
  The Visual Vertigo Analog Scale (VVAS) is a nine-item analog scale rating the level of symptoms provoked by daily situations typically inducing visual vertigo.

CONTACTS AND LOCATIONS:
Overall Officials: Russell Gore, MD, Principal Investigator — Sports Concussion Institute; David W Wright, MD, Principal Investigator — Emory University
Locations (1):
- Sports Concussion Institute, Atlanta, Georgia, United States